CLINICAL TRIAL: NCT00131053
Title: Phase 2 Study of Applying Pediatric Regimens to Younger Adult Patients With BCR-ABL-Negative Acute Lymphoblastic Leukemia
Brief Title: Applying Pediatric Regimens to Younger Adult Patients With Acute Lymphoblastic Leukemia (ALL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Adult Leukemia Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JALSG ALL202-U
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Lymphoblastic Leukemia, Acute
Keywords: acute lymphoblastic leukemia; newly diagnosed; BCR-ABL-negative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Methotrexate; Prednisolone; Dexamethasone; Vincristine; pirarubicin; Cyclophosphamide; Asparaginase; Cytarabine; Hydrocortisone; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Methotrexate; Drug: Prednisolone; Drug: Dexamethasone; Drug: Vincristine; Drug: Pirarubicin; Drug: Cyclophosphamide; Drug: L-asparaginase; Drug: Cytarabine; Drug: Hydrocortisone; Drug: Mercaptopurine

INTERVENTIONS:
Drug: Methotrexate
Drug: Prednisolone
Drug: Dexamethasone
Drug: Vincristine
Drug: Pirarubicin
Drug: Cyclophosphamide
Drug: L-asparaginase
Drug: Cytarabine
Drug: Hydrocortisone
Drug: Mercaptopurine

SUMMARY:
The purpose of this study is to investigate the efficacy and safety for treating adult ALL patients with the pediatric protocol.

DETAILED DESCRIPTION:
The prognosis for adult acute lymphoblastic leukemia (ALL) remains poor, which contrasts with that for pediatric ALL. It is regarded that the prognostic diversity is attributable to several differences between adults and children with respect to biological characteristics of leukemic cells, tolerance to anticancer drugs, treatment itself, and so on. It has been reported that adolescent ALL patients who were treated according to the pediatric protocol had a significantly better survival than those who were treated according to the adult protocol, indicating that the difference of treatment may be of considerable importance. To test the hypothesis, the Japan Adult Leukemia Study Group (JALSG) has planned a phase 2 study to treat younger ALL patients who are negative for BCR-ABL with the pediatric regimen which was used by the Japan Association of Childhood Leukemia Study. Those who are positive for BCR-ABL can participate in a separate protocol. The regimen is especially characterized by dose-intensified L-asparaginase, high-dose methotrexate, and intensified maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated BCR-ABL-negative ALL
* Age between 15 and 24 years
* Performance status between 0 and 3 (ECOG criteria)
* Adequate functioning of the liver (serum bilirubin level < 2.0 mg/dL); kidneys (serum creatinine level < 2.0 mg/dL); and heart (left ventricular ejection fraction greater than 50% and no severe abnormalities detected on electrocardiograms and echocardiographs).
* Written informed consent to participate in the trial

Exclusion Criteria:

* Uncontrolled active infection
* Another severe and/or life-threatening disease
* Positive for HIV antibody and/or hepatitis B surface (HBs) antigen tests
* Another primary malignancy which is clinically active and/or requires medical interventions
* Pregnant and/or lactating women
* Past history of renal failure

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-09; Primary Completion 2011-05 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
The rate of complete remission | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fumihiko Hayakawa, MD, Study Director — Nagoya University; Tomoki Naoe, MD, Study Chair — Nagoya University
Locations (1):
- Department of Hematology, Nagoya University Graduate School of Medicine, Nagoya, Japan

REFERENCES:
- See also: The JALSG homepage — http://www.jalsg.jp/